CLINICAL TRIAL: NCT05118516
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ASC43F, a Fixed-dose Combination (FDC) Oral Tablet Containing ASC41, a THR β Agonist and ASC42, an FXR Agonist in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of ASC43F, a Fixed Dose Combination Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASC43F-101
Record Dates: First submitted 2021-10-31; First posted 2021-11-12 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteer
Keywords: ASC43F; Phase 1; Thyroid hormone receptor beta agonist; FXR agonist; ASC41; ASC42

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): ASC43F for all subjects under the fasted state.
  Interventions: Drug: ASC43F

INTERVENTIONS:
Drug: ASC43F — One dose of oral ASC43F FDC tablet containing ASC41 5mg and ASC42 15mg.

SUMMARY:
This is a phase 1, open-label study in healthy adults. This study is aimed at evaluating the safety, tolerability, and pharmacokinetics of ASC43F, a fixed-dose combination (FDC) and single dose tablet containing ASC41, a THR β agonist and ASC42, an FXR agonist in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 to 65 years of age.
* Subjects must weigh at least 50 kg (110 pounds [lbs.]) for men, and at least 45 kg (99 lbs.) for women and body mass index (BMI) within the range 18.5-32 kilogram per meter square (kg/m2).
* Physical examination and vital signs are within normal range or slightly abnormal.

Exclusion Criteria:

* Any surgical or medical condition which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism, or excretion of drugs.
* Abnormal clinical or laboratory findings that indicate diseases including but not limited to renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic disease.
* History or current electrocardiogram (ECG) abnormalities, arrhythmias or heart valve diseases.
* History of viral hepatitis or HIV
* History of drug or food allergies that caused severe hypersensitivity reactions or anaphylaxis.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ASC43F evaluated by incidence of treatment emergent adverse events (TEAEs). | Baseline to day 7

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics as assessed by Cmax (Max Concentration) of ASC43F tablet following a single fixed oral dose in healthy subjects | Baseline to day 4
To evaluate the pharmacokinetics as assessed by Area Under the Curve (AUC) of ASC43F tablet following a single fixed oral dose in healthy subjects | Baseline to day 4
To evaluate the pharmacokinetics as assessed by Tmax (Time to Max Concentration) of ASC43F tablet following a single fixed oral dose in healthy subjects | Baseline to day 4

CONTACTS AND LOCATIONS:
Locations (1):
- 8307 Gault Lane, San Antonio, Texas, United States